CLINICAL TRIAL: NCT01273142
Title: A Prospective, Open-label 96-week Observational Pilot Study to Compare the Safety of Efavirenz Versus Nevirapine (Each in Combination With Zidovudine and Lamivudine or Tenofovir and Lamivudine) in Treating HIV Positive Patients With Mild Baseline Liver Function Test Impairment, and/or Hepatitis B or Hepatitis C Co-infection.
Brief Title: Compare to the Safety of Efavirenz and Nevirapine in Treating HIV Positive Patients With Mild Baseline Liver Function Test Impairment, and/or Hepatitis B or Hepatitis C Co-infection
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Henan Provincial People's Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Henan Provincial Hospital, Henan Provincial Infectious Disease Hospital
Other Study IDs: zzly-37183
Record Dates: First submitted 2011-01-06; First posted 2011-01-10 (Estimated); Last update posted 2011-01-10 (Estimated); Status verified 2010-12

CONDITIONS: HIV Infections; Liver Toxicity; Hepatitis Co-infection
Keywords: Human Immunodeficiency Virus, liver toxicity, hapatitis co-infection
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to demonstrate the difference in frequency and level of liver function disturbance between patients on efavirenz based ART, and patients on nevirapine based ART in HBV and HCV co-infected patients, (and/or with patients with abnormal liver function prior to ART), in China. Liver function tests will be measured at baseline and follow-up.

DETAILED DESCRIPTION:
The introduction of highly active antiretroviral therapy (HAART) has led to a significant reduction in AIDS-related morbidity and mortality. However, the frequent occurrence of chronic hepatitis progressing toward cirrhosis and/or hepatocarcinoma has been recognized as an increasing contributor to death of HIV-infected patients since early in the HAART era In China among the estimated 700,000 people living with HIV in China as of 20061, the percentage of HIV/HCV co-infected patients is high at 56.9%2. For these reasons, during HAART scrupulous attention should paid to the patients' liver function. At present, for price consideration, the NNRTI HIV drug used for antiretroviral therapy in China is nevirapine, which may lead to higher potential risk of liver function disturbance in clinical practice than efavirenz4-5.Roberto Manfredi and his colleagues3found that in a NVP treated group, patients showed at least a 2-fold increase of transaminases versus baseline as hepotoxicity index, while in EFV group, the number of patients with hepotoxicity showed a reduction, Also in the same study, time to reach transaminase peak value was shorter in the NVP group, which also demonstrate the liver toxicity side effect in NVP group. Recently some data has also shown an unusually high incidence of liver function disturbance in patients on HIV antiretroviral therapy in China6. Therefore to evaluate frequency and risk of patient hepatotoxicity caused by different HAART regimens in HBV-/HCV- co-infected HIV patients is necessary to provide evidence therapy for what HAART treatment should be used in China.

ELIGIBILITY:
Inclusion Criteria:

(Patients must meet all of the following criteria to enter this study.)

* Patients must be >18years of age and < 60 years of age
* Patients must be antiretroviral naive and have a HIV-1 RNA level≥500 copies/ml
* Patients with AST or ALT > 2x the upper limit of normal, and TBIL > 1.5x the upper limit of normal
* CD4 count to be <250 in female patients and <350 in male patients at entry
* Hemoglobin content to be > 90g/L
* Neutrophil cell count to be > 0.75 x 109/L
* Patients must be willing to accept the

Exclusion criteria:

(Patients meeting one or more of the following criteria will not be enrolled in this study.)

* Patients with allergies to or other contraindications for the selected ARV regimens.
* AST or ALT > 5x the upper limit of normal
* TBIL>2.5 x the upper limit of normal
* TB co-infection and other co-infection
* Pregnant or breastfeeding women
* Intravenous drug users
* Patient's education level that would interfere with the medical, adherence and withdrawal symptoms evaluation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Antiretroviral treatment naive patients with HIV-1 RNA level≥500 copies/ml and with AST or ALT > 2x the upper limit of normal, and TBIL > 1.5x the upper limit of normal.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-10 (Estimated); Study Completion 2012-12 (Estimated)